CLINICAL TRIAL: NCT00073580
Title: Angiomax in Patients With HIT/HITTS Type II Undergoing Off-PUMP CABG
Brief Title: Angiomax in Patients With HIT/HITTS Type II Undergoing Off-Pump Coronary Artery Bypass Grafting (CABG) (CHOOSE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC-BIV-02-02; CHOOSE
Record Dates: First submitted 2003-11-26; First posted 2003-11-27 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Thrombocytopenia; Thrombosis; Cardiac Disease; Coronary Artery Bypass Surgery
Keywords: HIT; HITTS; Heparin-antibodies; Coronary artery bypass surgery; CABG; Heparin-induced thrombocytopenia; Heparin-induced thrombocytopenia and thrombosis syndrome
MeSH Terms: conditions — Thrombocytopenia; Thrombosis; Heart Diseases | interventions — bivalirudin; Anticoagulants

INTERVENTIONS:
Drug: Angiomax (bivalirudin) anticoagulant — ): 250 mg vial administered as 0.75 mg/kg intravenous (IV) bolus and 1.75 mg/kg/h IV infusion for the duration of the procedure with the option to increase or decrease the infusion rate in 0.25 mg/kg/h increments or to administer additional 0.1-0.5 mg/kg boluses to maintain an activated clotting time (ACT+) >300 seconds. A low-dose infusion could be administered in the preoperative phase (up to 48 hours before the procedure) and in the postoperative phase (up to 14 days after the procedure) as clinically indicated for management of HIT/TS. An initial dose of 0.1 mg/kg IV bolus followed by an IV infusion of 0.2 mg/kg/h titrated to a desired activated partial thromboplastin time (aPTT), eg, 1.5-2.5 times baseline aPTT, was recommended.
  Other Names: bivalirudin

SUMMARY:
The purpose of this study is to examine the safety and efficacy of Angiomax as an anticoagulation in patients with heparin-induced thrombocytopenia (HIT)/heparin-induced thrombocytopenia with thrombosis syndrome (HITTS) undergoing off-pump coronary artery bypass (OPCAB) surgery.

ELIGIBILITY:
Inclusion:

* Be at least 18 years of age.
* Be accepted for OPCAB graft surgery (repeat CABG eligible)
* New diagnosis or history of objectively documented HIT/HITTS Type II, defined as:

  1. Positive heparin-induced platelet aggregation (HIPA) or other functional assay for HIT or immunoassay for HIT antibodies (ELISA), AND/OR
  2. HIT: Thrombocytopenia associated with heparin therapy, where the platelet count has decreased by 50%, OR
  3. HITTS: Thrombocytopenia (as defined in B above) PLUS any arterial or venous thrombosis (Deep-vein thrombosis, pulmonary embolism, mesenteric venouse or arterial thrombosis, acute myocardial infarction, left ventricular thrombus, ischemic stroke, or occlusion of limb arteries) diagnosed by physical exam/lab evidence and/or appropriate imaging studies (duplex ultrasound, venography, ventilation-perfusion scan, venouse or arterial angiography, MRI/MRA, catheterization.)

Exclusion Criteria:

* Confirmed pregnancy, by urine or serum pregnancy test (if woman of child-bearing potential).
* Cerebrovascular accident within 6 months, or any cerebrovascular accident with a residual neurological deficit.
* Intracranial neoplasm, arteriovenous malformation, or aneurysm.
* Dependency on renal dialysis or creatinine clearance <30mL/min.
* Ongoing treatment with warfarin (or other oral anticoagulant) at the time of enrollment.

Patients previously treated with warfarin may be enrolled if warfarin therapy can be safely discontinued and baseline INR is < 1.3 times control in the absence of heparin therapy.

* Known allergy to Angiomax or hirudin derived drugs, or known sensitivity to any component of the product.
* Patients receiving clopidogrel (Plavix®) within the previous 5 days may be enrolled if in the opinion of the Investigator the benefits of surgery outweigh the risk associated with recent clopidogrel administration.
* Patients receiving a glycoprotein IIb/IIIa inhibitor within the previous 48 hours if abciximab (ReoPro®) or 12 hours if eptifibatide (Integrilin®) or tirofiban (Aggrastat®), may be enrolled if in the opinion of the investigator the benefits of surgery outweigh the risk associated with not waiting the 48 or 12 hour time period prior to enrollment.
* Patients receiving lepirudin (Refludan®) or argatroban within the previous 24 hours prior to enrollment. Patients currently receiving lepirudin or argatroban can be enrolled if they are switched to Angiomax at least 24 hours prior to the contemplated OPCAB.
* Patients receiving low molecular weight heparin (LMWH) or thrombolytics within the previous 12 hours may be enrolled if in the opinion of the Investigator the benefits of surgery outweigh the risk associated with not waiting the 12 hour time period.
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of randomization.
* Refusal to undergo blood transfusion should it become necessary.
* Any other disease or condition, which, in the judgment of the investigator would place a patient at undue risk by being enrolled in the trial or inability to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2003-10; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | 7 days
  : In-hospital acute procedural success, defined as the absence of death, Q wave myocardial infarction (MI), repeat coronary revascularization, and stroke (hemorrhagic or ischemic) at hospital discharge or Day 7 after surgery ('Day 7/discharge'), whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Toval Rothschild, Ph.D., Study Director — The Medicines Company
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States